CLINICAL TRIAL: NCT00181298
Title: Memantine in Systemic Lupus Erythematosus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Dr. Michelle Petri, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAM-MD-20
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2008-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Memantine; SLE; Anti NR2; ANAM; Cognitive functioning
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Memantine
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — Dispensing initially 5 mg. Dose Increased by 5 mg weekly to 20 mg/d final dose by week 4.
  Other Names: Namenda
  Arms: 1
Drug: Placebo — Dispensing initially 5 mg. Dose Increased by 5 mg weekly to 20 mg/d final dose by week 4
  Arms: 2

SUMMARY:
Neuropsychiatric manifestations of Systemic Lupus Erythematosus (NPSLE) are both common and an important source of morbidity. Of the case definitions for NPSLE syndromes that have recently been developed, cognitive dysfunction appears to be the most prevalent. A novel mechanism is that a subset of SLE patients with cognitive dysfunction have antibodies in the NR2 glutamate receptor. We propose, in a double -blind placebo-controlled trial, to determine whether SLE patients, with or without the NR2 glutamate receptor antibody, have significant improvement using memantine, an inhibitor of the NMDA receptor.

DETAILED DESCRIPTION:
Patients with SLE frequently report cognitive and memory problems and many studies have documented significant cognitive deficits with traditional neuropsychological test batteries. Many traditional neuropsychological tests are unsuitable for repeated measures over short intervals caused by expected improvement due to test-retest or practice effects. We will utilize an automated battery (ANAM) of cognitive function tests at baseline, 6 weeks, and 12 weeks, as the outcome measure.

Betty Diamond M.D. and colleagues demonstrated that a subset of lupus anti-DNA antibodies cross-reacts with the NR2 glutamate receptor in patients with SLE. Glutamate receptors can display altered expression in major psychosis and over-stimulation of NR2 can cause excitotoxic neuron death through excessive entry of calcium into cells. Thus, antibody reactivity with NR2a or NR2b may not only serve as a marker for CNS disease in SLE but may also be neuropathogenic mechanism for some of the non-focal CNS disturbances in SLE.

Memantine is a low- to moderate-affinity, noncompetitive N-methyl-D-asparate (NMDA) receptor that represents the first member of a new class of medications showing clinical benefit and good tolerability in Alzheimer's Disease. Because of our anecdotal experience with some SLE patients with cognitive impairment improving with donepezil therapy, an approved Alzheimer's Disease therapy, and because of the known association of cognitive impairment in SLE with anti-NR2 glutamate (NMDA) receptor antibodies, we hypothesize that memantine will have benefit for cognitive dysfunction in SLE.

We believe that computerized cognitive function batteries (ANAM) can be used in clinical trials of cognitive impairment, with the benefit of efficiency, immediate results, and less patient time. However, because this is the first clinical trial of this kind in SLE, we will also use the formal American College of Rheumatology neuropsychiatric battery, as well

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of SLE
* Self-reported cognitive impairment

Exclusion Criteria:

* Age < 18 years.
* History of non-compliance
* Pregnancy
* Liver or renal insufficiency/failure (calculated creatinine clearance < 50 cc/min)
* Severe SLE flare in the last 6 weeks (defined as SLEDAI > 12 points)
* Recent (within 4 weeks) change in any medication relevant to cognitive function, including prednisone, anti-depressants, medications for insomnia, narcotic medications, attention deficit disorder medications
* Current alcohol or illicit drug abuse
* Current use of Namenda, Aricept, Provigil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2006-03; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Change in ANAM, Version 3.11 | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Petri, M.D., M.P.H., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Lupus Center, 1830 East Monument Street, Suite 7500, Baltimore, Maryland, United States